CLINICAL TRIAL: NCT07312877
Title: Comparison of the Effectiveness of Intraoperative Intravenous Lidocaine and Intravenous Remifentanil in Postoperative Pain Management in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Nilsu GÜNDÜZ, resident doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: NG269436444.
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Colicystitis
MeSH Terms: interventions — Lidocaine; Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lidocaine Group: Patients received IV lidocaine (1 mg/kg bolus + infusion) during laparoscopic cholecystectomy
  Interventions: Drug: Lidocaine
- Remifentanil Group: Patients received IV remifentanil infusion during laparoscopic cholecystectomy
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Lidocaine — Patients received intravenous lidocaine 1 mg/kg bolus followed by continuous infusion during laparoscopic cholecystectomy.
  Groups: Lidocaine Group
Drug: Remifentanil — Patients received intravenous remifentanil infusion during laparoscopic cholecystectomy.
  Groups: Remifentanil Group

SUMMARY:
This study aims to compare the effects of intraoperative intravenous lidocaine and intravenous remifentanil on postoperative pain management in patients undergoing laparoscopic cholecystectomy under general anesthesia. Although laparoscopic procedures are minimally invasive, patients frequently experience postoperative pain. Multimodal analgesia techniques are recommended to optimize pain control and recovery while minimizing opioid-related adverse effects.

In this prospective observational study, adult patients (ASA I-II) aged over 18 years who provided written informed consent were included. Standard intraoperative monitoring was performed. Anesthesia induction consisted of fentanyl, lidocaine, propofol, and rocuronium, with maintenance using sevoflurane. Hemodynamic parameters were recorded throughout the procedure. For postoperative analgesia, intravenous paracetamol and tramadol were administered before the end of anesthesia.

The primary objective is to evaluate whether intravenous lidocaine provides postoperative analgesic efficacy and recovery quality comparable to remifentanil, and to determine its potential role as an opioid-sparing alternative in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This prospective observational study was designed to compare the effects of intraoperative intravenous lidocaine and intravenous remifentanil on postoperative pain control, hemodynamic stability, and recovery quality in patients undergoing elective laparoscopic cholecystectomy under general anesthesia. Although laparoscopic surgery is minimally invasive, patients frequently experience moderate to severe postoperative pain, which can delay recovery and discharge. Multimodal analgesia strategies have been developed to improve postoperative comfort while minimizing the adverse effects of opioids such as respiratory depression, nausea, and delayed recovery.

The study was conducted following approval from the institutional ethics committee, and written informed consent was obtained from all participants. Patients aged over 18 years with an ASA physical status of I-II were included. Standard monitoring (DII and V5 ECG, non-invasive blood pressure, and pulse oximetry) was applied upon arrival in the operating room. General anesthesia was induced with fentanyl (1-2 mcg/kg), lidocaine (1 mg/kg), propofol (2-2.5 mg/kg), and rocuronium (0.6 mg/kg). Anesthesia was maintained with sevoflurane in oxygen/air mixture.

Hemodynamic parameters, including heart rate, systolic, diastolic, and mean arterial pressures, and oxygen saturation (SpO₂), were recorded at baseline and at defined intraoperative intervals. Twenty minutes before the end of the procedure, intravenous paracetamol (15 mg/kg) and tramadol hydrochloride (10 mg/kg) were administered for postoperative analgesia. After emergence from anesthesia, patients were transferred to the post-anesthesia care unit (PACU) and then to the ward once the Aldrete recovery score reached 9.

Postoperative pain intensity was assessed using the Numeric Rating Scale (NRS) at regular intervals for 24 hours. When NRS > 4, rescue analgesia was administered according to the institutional protocol. The collected data were analyzed to compare intraoperative hemodynamic stability, depth of anesthesia, postoperative recovery characteristics, and analgesic requirements between the lidocaine and remifentanil groups.

The primary hypothesis of this study is that intravenous lidocaine can provide comparable postoperative analgesia to remifentanil, with potential benefits such as improved hemodynamic stability, faster recovery, and fewer opioid-related side effects. The findings may support the use of lidocaine as an effective opioid-sparing alternative in multimodal analgesia protocols for laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* ASA physical status I-II
* Scheduled for elective laparoscopic cholecystectomy under general anesthesia
* Provided written and verbal informed consent

Exclusion Criteria:

* Allergy or contraindication to lidocaine, remifentanil, or study drugs
* Severe cardiovascular, hepatic, or renal disease
* Pregnancy or lactation
* Conversion from laparoscopic to open cholecystectomy
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (ASA I-II) undergoing elective laparoscopic cholecystectomy under general anesthesia at Prof. Dr. Cemil Taşçıoğlu City Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score (NRS) | Within 24 hours after surgery
  Postoperative pain intensity will be assessed using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst pain imaginable). Pain scores will be recorded at rest at 1, 6, 12, and 24 hours after surgery. The comparison between the lidocaine and remifentanil groups will determine the effect of intraoperative intravenous lidocaine versus remifentanil on postoperative analgesia.

SECONDARY OUTCOMES:
Heart Rate | Intraoperative period
  Changes in heart rate will be recorded at baseline, during pneumoperitoneum, and throughout surgery to evaluate intraoperative hemodynamic stability between groups.
Mean Arterial Pressure | Intraoperative period
  Changes in mean arterial blood pressure will be recorded at baseline, during pneumoperitoneum, and throughout surgery to evaluate intraoperative hemodynamic stability between groups.
Systolic Blood Pressure | Intraoperative period
  Changes in systolic blood pressure will be recorded at baseline, during pneumoperitoneum, and throughout surgery to evaluate intraoperative hemodynamic stability between groups.
Diastolic blood Pressure | Intraoperative period
  Changes in diastolic blood pressure will be recorded at baseline, during pneumoperitoneum, and throughout surgery to evaluate intraoperative hemodynamic stability between groups.
Recovery Profile | Immediate postoperative period
  Time to reach an Aldrete score ≥9 (range 0-10, with higher scores indicating better recovery) will be measured to evaluate the effect of intraoperative lidocaine versus remifentanil on recovery characteristics.
Postoperative Analgesic Requirement | First 24 hours postoperatively
  Total amount of rescue analgesic medication administered (tramadol and paracetamol) within 24 hours after surgery will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascıoğlu City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No